CLINICAL TRIAL: NCT03290365
Title: The Combination Long-term Effect of Platelet-rich Plasma and Hyaluronic Acid in Patients With Knee Osteoarthritis: a Prospective Randomized Double-blind Controlled Trial
Brief Title: The Combination Effect of Platelet-rich Plasma and Hyaluronic Acid for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP and HA for OA knee
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Knee Osteoarthritis
Keywords: Platelet rich plasma; Osteoarthritis of knee; Hyaluronic acid
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet rich plasma + Hyaluronic acid (Active Comparator): Platelet rich plasma (PRP) and Hyaluronic acid (HA) are beneficial for patients with osteoarthritis of knee. Patients received one dose of PRP injection. One week later, the one dose of HA is injected for intervention group.
  Interventions: Drug: platelet rich plasma + Hyaluronic acid
- Platelet rich plasma + normal saline (Placebo Comparator): Patients received one dose of PRP injection. One week later, the one dose of normal saline is injected for control group.
  Interventions: Drug: platelet rich plasma + normal saline

INTERVENTIONS:
Drug: platelet rich plasma + Hyaluronic acid — Platelet rich plasma (PRP) and Hyaluronic acid (HA) are beneficial for patients with osteoarthritis of knee.
  Arms: Platelet rich plasma + Hyaluronic acid
Drug: platelet rich plasma + normal saline — The normal salin as the placebo intervention was injection control group.
  Arms: Platelet rich plasma + normal saline

SUMMARY:
Although platelet rich plasma (PRP) and Hyaluronic acid (HA) are beneficial for osteoarthritis of knee (OA knee), the combined effect of PRP with HA was not clear so far. Hence, investigator assess a prospective randomized double-blind controlled trial.

DETAILED DESCRIPTION:
Patients with single or bilateral OA knee will be enrolled and randomized into intervention and control group. One dose of PRP is applied into both groups. One week later, one dose of HA is injected in intervention group and one dose of normal saline is injected in control group. Outcome measurements included visual analog scale (VAS)、Lequesne's severity index、Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)、balance test (Biodex) and analysis of synovial fluid at different follow-up frame (1st month, 3rd month, 6th month and 1 year after treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50 to 75 y/o.
2. Alert consciousness
3. Symptom of knee osteoarthritis persist at least 6 months and stage I to III scored by Ahlbäck grading system
4. The pain score measured by VAS at least 4 points

Exclusion Criteria:

1. Has received hyaluronic acid, PRP or steroid injection within 6 months
2. Has received NSAIDs or steroid within one week
3. Tumor or metastasis surrounding the knee joint
4. Has received total knee replacement, major surgery in knee, rheumatoid arthritis
5. Patient who cant tolerance the balance test.
6. Thrombocytopenia or coagulopathy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in severity of symptoms and functional status on 1st month, 3rd month, 6th month and one year after injection. | Pre-treatment, 1st month, 3rd month, 6th month and one year after injection.
  Using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) to measure the symptoms and functional status before treatment and multiple time frame after treatment. Both subscales has the scores ranged from 1 to 5 for each item and a higher score indicating more severe of symptom or impaired functional status.

SECONDARY OUTCOMES:
Change from baseline in severity of symptoms and functional status on 1st month, 3rd month, 6th month and one year after injection. | Pre-treatment, 1st month, 3rd month, 6th month and one year after injection.
  Using the Lequesne's severity index to measure the symptoms and functional status before treatment and multiple time frame after treatment. A higher score indicate more severe.
Change from baseline of pain on 1st month, 3rd month, 6th month and one year after injection. | Pre-treatment, 1st month, 3rd month, 6th month and one year after injection.
  Using the Visual analog scale (VAS) to measure the pain scale before treatment and multiple time frame after treatment. The score ranging from 10 (remarkable pain) to 0 (no pain).
Change from baseline in balance function on 1st month, 3rd month, 6th month and one year after injection. | Pre-treatment, 1st month, 3rd month, 6th month and one year after injection.
  Using the balance test (Biodex) to measure the balance function before treatment and multiple time frame after treatment.
Change from baseline in analysis of synovial fluid on 6th month and one year after injection. | Pre-treatment, 6th month and one year after injection.
  The synovial fluid is aspirated to measure the parameters before treatment and multiple time frame after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, National Defense Medical Center
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

REFERENCES:
- [Result] Abate M, Verna S, Schiavone C, Di Gregorio P, Salini V. Efficacy and safety profile of a compound composed of platelet-rich plasma and hyaluronic acid in the treatment for knee osteoarthritis (preliminary results). Eur J Orthop Surg Traumatol. 2015 Dec;25(8):1321-6. doi: 10.1007/s00590-015-1693-3. Epub 2015 Sep 24. PMID 26403468
- [Result] Lana JF, Weglein A, Sampson SE, Vicente EF, Huber SC, Souza CV, Ambach MA, Vincent H, Urban-Paffaro A, Onodera CM, Annichino-Bizzacchi JM, Santana MH, Belangero WD. Randomized controlled trial comparing hyaluronic acid, platelet-rich plasma and the combination of both in the treatment of mild and moderate osteoarthritis of the knee. J Stem Cells Regen Med. 2016 Nov 29;12(2):69-78. doi: 10.46582/jsrm.1202011. eCollection 2016. PMID 28096631
- [Result] Chen SH, Kuan TS, Kao MJ, Wu WT, Chou LW. Clinical effectiveness in severe knee osteoarthritis after intra-articular platelet-rich plasma therapy in association with hyaluronic acid injection: three case reports. Clin Interv Aging. 2016 Sep 8;11:1213-1219. doi: 10.2147/CIA.S114795. eCollection 2016. PMID 27660427
- [Result] Dallari D, Stagni C, Rani N, Sabbioni G, Pelotti P, Torricelli P, Tschon M, Giavaresi G. Ultrasound-Guided Injection of Platelet-Rich Plasma and Hyaluronic Acid, Separately and in Combination, for Hip Osteoarthritis: A Randomized Controlled Study. Am J Sports Med. 2016 Mar;44(3):664-71. doi: 10.1177/0363546515620383. Epub 2016 Jan 21. PMID 26797697